CLINICAL TRIAL: NCT05298462
Title: Clinical Evaluation of Rapid Antibody Test for Covid-19
Acronym: CERAbTc-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: West Hertfordshire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 56480; 283264 (Other: IRAS)
Record Dates: First submitted 2022-03-25; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In this study we aim to evaluate the accuracy of this new test, in patients and in hospital staff with a history of COVID-19 symptoms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other)
  Interventions: Diagnostic Test: Livzon Rapid Antibody Test for COVID-19
- Hospital staff (Other)
  Interventions: Diagnostic Test: Livzon Rapid Antibody Test for COVID-19

INTERVENTIONS:
Diagnostic Test: Livzon Rapid Antibody Test for COVID-19 — Point-of-care Rapid Antibody Test for COVID-19

SUMMARY:
Rapid, accurate diagnosis of Covid-19 would greatly help to improve clinical management of patients presenting with symptoms of possible Covid-19. Currently results of the standard test for the virus take 2-3 days to be reported.

Watford General Hospital has imported rapid antibody tests manufactured by Zuhai Livzon Diagnostics Inc in China and our team would like to evaluate their accuracy and clinical usefulness. The test involves taking a drop of blood from the patient (either from a venous blood sample taken for other blood tests, or from a fingerprick). This is applied to a test strip (similar to a pregnancy test) and two drops of diluent are added. If the patient has antibodies to Covid-19, two lines appear on the test strip (like a positive pregnancy test) whereas if the patient has no antibodies, only one line appears (like a negative pregnancy test). There are two different types of antibody: IgM is produced early in the course of the illness (day 7-14) and then IgG is produced later and continues to be present, probably for months or years. There are two test strips, one for each of these types of antibody.

In this study we aim to evaluate the accuracy of this new test, in three groups of patients. Firstly those with proven Covid-19 and at least 7 days after the onset of their illness. We aim to recruit 200 patients in total: at least 138 patients with 10 or more days of symptoms, plus a subgroup of up to 62 patients with 7-9 days of symptoms (to explore the usefulness of the test earlier in the course of illness). The second group of 250 patients will be those hospital staff who report symptoms possibly caused by Covid-19 and are receiving a standard antibody test.

The third group of patients will be those followed up in a "virtual hospital" for clinically suspected Covid-19 who had never been tested with a standard PCR test.

As we are not sure of the accuracy of the new test, its results will not be used to make decisions about treatment for the patient.

This study will enable us to discover rapidly whether the new test is accurate, and if so we will conduct further studies to assess how it can help to improve management of patients with suspected Covid-19.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient or patient in the "virtual hospital" with confirmed Covid-19 infection on PCR OR with history of clinically suspected Covid-19 but no PCR test OR hospital staff with clinical suspicion of past Covid-19 infection.
2. Age 18 or over
3. At least 7 days since onset of symptoms
4. Willing and able to give written informed consent

Exclusion Criteria:

1. Symptom duration <7 days.
2. Lack of written consent
3. Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2020-05-17 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | At least 7 days after onset of symptoms
  Sensitivity and specificity compared to standard PCR and/or venous antibody test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Moore, FRCGP, Principal Investigator — University of Southampton
Locations (1):
- Watford General Hospital, Watford, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vancheeswaran R, Willcox ML, Stuart B, Knight M, Kandil H, Barlow A, Patel MH, Stockham J, O'Neill A, Clark TW, Wilkinson T, Little P, Francis N, Griffiths G, Moore M. Accuracy of rapid point-of-care antibody test in patients with suspected or confirmed COVID-19. J Infect. 2022 Jan;84(1):94-118. doi: 10.1016/j.jinf.2021.07.006. Epub 2021 Jul 14. No abstract available. PMID 34273411
- See also: Pre-print — https://www.medrxiv.org/content/10.1101/2020.11.17.20233296v1